CLINICAL TRIAL: NCT02639156
Title: Evaluation of Tolerance and Acceptability of AYMES 'LONDON' Product
Brief Title: Acceptability and Tolerance of New Oral Nutritional Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aymes International Limited (Industry)
Collaborators: Alison Clark Health and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AY:SPT1
Record Dates: First submitted 2015-12-18; First posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-08

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention (Experimental): Patients established on an oral nutritional supplement, being prescribed 1-2 ONS providing at least 300kcal/day will be changed onto an equivalent prescription of AYMES LONDON for a period of 9 days.
  Interventions: Dietary Supplement: AYMES LONDON

INTERVENTIONS:
Dietary Supplement: AYMES LONDON — AYMES LONDON is a powder, designed to be mixed with 75ml whole milk to make a dessert style ONS. When made-up, AYMES LONDON provides 303kcal (2.2kcal/ml) and 11.2g protein. It is not designed to be used as a sole source of nutrition. It is a Food for Special Medical Purposes (FSMP) and must therefore be used under medical supervision.

SUMMARY:
To evaluate tolerance and acceptability of AYMES LONDON in patients requiring supplementary oral nutritional support compared with currently available alternatives.

DETAILED DESCRIPTION:
TITLE EVALUATION OF TOLERANCE AND ACCEPTABILITY OF AYMES LONDON STUDY OBJECTIVES

* To evaluate tolerance and acceptability of AYMES LONDON in patients requiring supplementary oral nutritional support compared with currently available alternatives.
* To obtain data to support an ACBS submissions for AYMES LONDON (to allow for prescription in the community at NHS expense).

STUDY DESIGN Interventional study. STUDY POPULATION 20 patients established on an oral nutritional supplement (ONS), requiring nutritional supplementation of at least 300kcal/day. Patients residing in community settings (e.g. own home, care home or community hospital) STUDY PRODUCTS AYMES LONDON Patients' current oral nutritional supplements STUDY GROUPS This is an observational study where the patient will act as their own control, there will be just one study group containing all patients STUDY OUTLINE Baseline: After recruitment patients will remain on their current oral nutritional supplement for 3 days, during which time baseline tolerance data will be recorded (number and consistency of bowel movements, daily, volume of ONS taken, any episodes of nausea, vomiting, burping, abdominal pain, bloating or diarrhoea). A three-day food diary will be kept to record total oral intake. Patients will also have anthropometric measurements carried out during this period (weight, height, body mass index (BMI)).

Intervention Period : Patients will then be changed onto an equivalent prescription of AYMES LONDON for a period of 9 days. Tolerance data will be recorded daily but the first 2 days on AYMES LONDON will be considered a 'transitional' period and data from these days will not be analysed. A further 3-day food diary will be kept during the intervention period. Weight of the patient will be recorded at the end of the period on AYMES LONDON, and an acceptability questionnaire will be completed.

Comparisons will be made between baseline and the end of each phase of the study using appropriate analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who are able to communicate their views regarding acceptability.
* Patients established on an oral nutritional supplement, being prescribed 1-2 ONS providing at least 300kcal/day
* Patients expected to require oral nutritional supplementation for at least 2 further weeks.
* Informed consent obtained

Exclusion Criteria:

* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study
* Patients requiring a milk free
* Patients with medical or dietary contraindication to any feed ingredients (see appendix 2 of protocol for full list)
* Patients with significant renal or hepatic impairment
* Patients with dysphagia requiring stage 1,2 or 3 thickened fluids
* Patients with uncontrolled inflammatory bowel disease or previous bowel resection with ongoing gastrointestinal symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
GI Side Effects when using AYMES LONDON | 9 days
  Recording of any nausea, vomiting, abdominal pain, bloating / flatulence when using AYMES LONDON as assessed by presence / absence of side effect compared to baseline period

SECONDARY OUTCOMES:
Change to bodyweight of subjects when using AYMES LONDON | 9 DAYS
  Recording of body weight (kg) at start of study, start of intervention and end of intervention for comparison to investigate any significant weight change during the intervention period when compared to baseline.
Compliance with prescription of AYMES LONDON | 9 days
  Recording of amount of AYMES LONDON consumed by subjects to be compared to amount prescribed of intervention period compared to baseline period.
Bowel habits of subjects when using AYMES LONDON | 9 days
  Recording of bowel habits for one week using AYMES LONDON (as assessed by frequency and consistency of bowel movements (assessed by Bristol Stool Scale for consistency, and frequency of bowels open) compared to baseline period.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Clark, BSc (Hons), Principal Investigator — Alison Clark Health and Nutrition

REFERENCES:
- [Background] Stratton RJ, Green CJ, Elia M. Disease-related malnutrition: an evidence based approach to treatment. Wallingford: CABI Publishing; 2003.
- [Background] National Institute for Health and Care Excellence (NICE). Nutrition support in adults: oral nutrition support, enteral tube feeding and parenteral nutrition (clinical guideline 32). 2006. London, National Institute for Health and Clinical Excellence (NICE).
- [Background] Stratton RJ, Elia M. A review of reviews: A new look at the evidence for oral nutritional supplements in clinical practice. Clin Nutr 2007; 2(Suppl 1):5-23.
- [Background] Gazzotti C, Arnaud-Battandier F, Parello M, Farine S, Seidel L, Albert A, Petermans J. Prevention of malnutrition in older people during and after hospitalisation: results from a randomised controlled clinical trial. Age Ageing. 2003 May;32(3):321-5. doi: 10.1093/ageing/32.3.321. PMID 12720620
- [Background] Manders M, de Groot CP, Blauw YH, Dhonukshe-Rutten RA, van Hoeckel-Prust L, Bindels JG, Siebelink E, van Staveren WA. Effect of a nutrient-enriched drink on dietary intake and nutritional status in institutionalised elderly. Eur J Clin Nutr. 2009 Oct;63(10):1241-50. doi: 10.1038/ejcn.2009.28. Epub 2009 May 20. PMID 19455176
- [Background] Wouters-Wesseling W, Wouters AE, Kleijer CN, Bindels JG, de Groot CP, van Staveren WA. Study of the effect of a liquid nutrition supplement on the nutritional status of psycho-geriatric nursing home patients. Eur J Clin Nutr. 2002 Mar;56(3):245-51. doi: 10.1038/sj.ejcn.1601319. PMID 11960300
- [Background] Hubbard GP, Elia M, Holdoway A, Stratton RJ. A systematic review of compliance to oral nutritional supplements. Clin Nutr. 2012 Jun;31(3):293-312. doi: 10.1016/j.clnu.2011.11.020. Epub 2012 Jan 17. PMID 22257636